CLINICAL TRIAL: NCT06700161
Title: Investigation of Lipoxin A4, Annexin A1 and Interleukin-1 Beta Levels in Gingival Crevicular Fluid in Individuals With Stage 3 Grade A Periodontitis
Brief Title: Investigation of Lipoxin A4, Annexin A1 and Interleukin-1 Beta Levels in Individuals With Periodontitis.
Acronym: Lipoxin A4
Status: Completed | Type: Observational
Sponsor: Eda Cetin Ozdemir (Other)
Responsible Party: Sponsor-Investigator, Eda Cetin Ozdemir, Principal Investigator, Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Other Study IDs: 09.05.2024-117; 2024/4-13 M (Other Grant/Funding Number: Scientific Research Projects Coordination Unit of Kahramanmaraş Sütçü İmam University)
Record Dates: First submitted 2024-11-15; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Peridontal Disease
Keywords: periodontal disease; Anneksin; lipoksin
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Healthy group
  Interventions: Other: Obtaining CGF from patients
- Test group: Stage III Grade C Periodontitis
  Interventions: Other: Obtaining CGF from patients

INTERVENTIONS:
Other: Obtaining CGF from patients — Periodontal clinical parameters and Annexin and Lipoxin parameters in CGF will be compared between the test and control groups

SUMMARY:
Since the researchers thought that Annexin A1, Lipoxin A4 and IL-1 Beta parameters, which have been found to be related to inflammatory conditions, may increase in periodontitis, a common inflammatory gum disease, we wanted to evaluate the changes in Annexin A1, Lipoxin A4 and IL-1 Beta levels in the Gingival Crevicular Fluid of participants with periodontitis.

DETAILED DESCRIPTION:
Periodontitis is a chronic, multifactorial inflammatory disease characterized by microbial-mediated, host-mediated inflammation, resulting in periodontal attachment loss and eventual tooth loss. Given the high prevalence and systemic effects of periodontitis, research into the pathogenesis and treatment of periodontal disease is crucial to improving oral health and overall health outcomes.

In recent years, there has been great interest in determining the role of lipid mediators in pro- and anti-inflammatory events, which are of great importance in the pathogenesis of periodontitis. LIPOXIN A4 (LXA4), which serves as an inflammatory shutdown signal, is produced from arachidonic acid via interactions between individual lipoxygenases. Preclinical models have demonstrated the potential and efficacy of LXA4 in preventing the onset of periodontitis and treating periodontal disease by regenerating lost periodontium. LXA4 is produced by the dual oxygenation of arachidonic acid by 5-lipoxygenase and 12-lipoxygenase and mediates inflammatory suppression signals in vivo. LXA4 is biosynthesized by leukocytes, endothelial cells, and platelets via transcellular pathways and has potent inhibitory effects on various inflammatory mechanisms.

Annexins (ANXA) belong to the calcium (Ca+2) binding protein family that plays a role in inflammatory host defense. ANXA1, also known as lipocortin 1, is an anti-phospholipase protein that binds to cell membranes via a calcium-dependent pathway. ANXA1 inhibits the production of proinflammatory lipid mediators by inhibiting the activity of phospholipase A2. In addition, ANXA1 can modify many different steps and various cells involved in the inflammatory process. ANXA1 has long been classified as an anti-inflammatory protein due to its control over leukocyte-mediated immune responses. An ex vivo study has shown that the induction and translocation of ANXA1 protein to the cell membrane is stimulated by IL-6 . It has also been reported to be a critical negative regulator of proinflammatory mediators including IL-1, IL-6 and cyclooxygenase-2, while it has also been reported to stimulate the release of the anti-inflammatory cytokine IL-10 .

Since the researchers thought that Annexin A1, Lipoxin A4 and IL-1 Beta parameters, which have been found to be related to inflammatory conditions, may increase in periodontitis, a common inflammatory gum disease, we wanted to evaluate the changes in Annexin A1, Lipoxin A4 and IL-1 Beta levels in the Gingival Crevicular Fluid of participants with periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be a volunteer
* He/she must be over 18 years old
* He/she must not have any systemic disease

Exclusion Criteria:

* Smoking, drinking alcohol
* Being pregnant or breastfeeding
* Not volunteering
* Having had periodontal treatment in the last 6 months
* Having used antibiotics or anti-inflammatory drugs in the last 6 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients applying to Kahramanmaraş Sütçü İmam University, Faculty of Dentistry, Department of Periodontics
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-03-16 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Changes in Annexin and Lipoxin parameters in CGF in periodontal disease | 6 mounth
  We expect Annexin and Lipoxin parameters to decrease and IL-1b levels to increase in periodontal disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Sütçü İmam University, Faculty of Dentistry, Department of Periodontics, Kahramanmaraş, Onikişubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
ı don't want to share

REFERENCES:
- [Background] Tobon-Arroyave SI, Isaza-Guzman DM, Gomez-Ortega J, Florez-Alzate AA. Salivary levels of specialized pro-resolving lipid mediators as indicators of periodontal health/disease status. J Clin Periodontol. 2019 Oct;46(10):978-990. doi: 10.1111/jcpe.13173. Epub 2019 Aug 20. PMID 31339183
- [Background] Casarin RCV, Salmon CR, Stolf CS, Paz HES, Rangel TP, Domingues RR, Pauletti BA, Paes-Leme AF, Araujo C, Santamaria MP, Ruiz KS, Monteiro MF. Salivary annexin A1: A candidate biomarker for periodontitis. J Clin Periodontol. 2023 Jul;50(7):942-951. doi: 10.1111/jcpe.13803. Epub 2023 Mar 19. PMID 36935103
- [Background] Ma R, Liu Y, Xu Y, Duan D. Lipoxin A4 levels predict site-specific clinical improvements post scaling and root planing and correlate negatively with periodontal pathogens in severe periodontitis. BMC Oral Health. 2024 Feb 8;24(1):204. doi: 10.1186/s12903-024-03948-w. PMID 38331747
- [Background] Schenkein HA, Papapanou PN, Genco R, Sanz M. Mechanisms underlying the association between periodontitis and atherosclerotic disease. Periodontol 2000. 2020 Jun;83(1):90-106. doi: 10.1111/prd.12304. PMID 32385879
- See also: Reference link to study protocol — https://pubmed.ncbi.nlm.nih.gov/36935103/
- Available data/document: Study Protocol: Study Protocol — https://tipfakultesi.ksu.edu.tr/Default.aspx?SId=24451